CLINICAL TRIAL: NCT03410589
Title: Desenvolvimento de Teste Adaptativo Computadorizado (CAT) Para avaliação do Sono, Fadiga e Qualidade de Vida em Pacientes Com Dor crônica
Brief Title: Development of a Computerized Adaptive Test (CAT) for Evaluation of Sleep, Fatigue and Quality of Life in Patients With Chronic Pain
Acronym: CAT
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, Principal Investigator, University of Sao Paulo
Other Study IDs: CAT
Record Dates: First submitted 2018-01-10; First posted 2018-01-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm
  Interventions: Other: Sinlge arm

INTERVENTIONS:
Other: Sinlge arm — application of scales for evaluation of sleep, fatigue and quality of life - Observational study

SUMMARY:
The purpose of this study is to evaluate quality of life, sleep and fadigue in patients with chronic pain using an Item-Response Theory methodology and also generating a Computer Adaptive Testing System

ELIGIBILITY:
Inclusion Criteria:

be able to read Portuguese be able to write Portuguese being in treatment for chronic pain

Exclusion Criteria:

hearing impairment that impairs ability to respond to tests visual impairment that impairs ability to respond to tests physical impairment that impairs ability to respond to tests cognitive impairment that impairs ability to respond to tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
sleep disorders | Within 1 month before the study start
  score in Pittsburgh Sleep Quality
fatigue | Within 7 days before the study start
  score of Multidimensional Fatigue Inventory
measurement quality of live | Within 1 month before the study start
  measurement quality of live will be score the using SF-12
sleep disorders | Within 1 month before the study start
  score Index and Insomnia Severity Index (ISI)
measurement quality of live | Within 1 month before the study start
  measurement quality of live will be WHOQOL-bref

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Andrade, PhD, Principal Investigator — doctor and investigator
Locations (1):
- Hospital das clinicas da FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided